CLINICAL TRIAL: NCT06713733
Title: Comparison of Clinical Efficacy of Submucosal Dexamethasone and Oral Trypsin-chymotrypsin for Reduction of Postoperative Sequelae After Lower Third Molar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, DR. SABIN BANIYA, DR.SABIN BANIYA, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRC/2765/024
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Clinical Efficacy of Submucosal Dexamethasone and Oral Trypsin Chymotrypsin for Reduction of Postoperative Sequelae After Lower Third Molar Surgery
Keywords: Dexamethasone; Trypsin-chymotrypsin
MeSH Terms: interventions — Dexamethasone; Chymotrypsin; chymotrypsin, trypsin drug combination

STUDY DESIGN:
Intervention Model Description: group a - submucosal dexamethasone group b - oral trypsin chymotrypsin
Who Masked: Investigator
Masking Description: PI does not have access to any of the groups. i.e PI is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): submucosal dexamethasone is quite simple, less invasive, painless, convenient for the surgeon and offers a low cost solution. Submucosal injection offers advantage of concentrating the drug near the surgical area with less systemic absorption and no further manipulation of the tissues.
  preoperative submucosal dexamethasone 8mg prior to incision locally.
  Interventions: Drug: Dexamethasone
- Chymotrypsin (Active Comparator): oral trypsin chymotrypsin is proteolytic enzymes.
  1 tab given 30 minutes prior to incision and 1 tab for three times a day for 5 days after extraction.
  Interventions: Drug: Chymotrypsin

INTERVENTIONS:
Drug: Dexamethasone — local infiltration
  Other Names: submucosal dexamethasone
  Arms: Dexamethasone
Drug: Chymotrypsin — orally given
  Other Names: oral trypsin chymotrypsin
  Arms: Chymotrypsin

SUMMARY:
Pain, edema and trismus are the most frequent postoperative sequelae to surgical removal of impacted teeth, all of are due to the local inflammatory response.

Use of corticosteroids decrease tissue mediators of inflammation and reduce edema.

Use of trypsin-chymotrypsin elaborates the enzymes esterase in blood plasma that inhibits inflammation by hydrolytic degradation of the inflammatory peptides.

DETAILED DESCRIPTION:
Impacted tooth is a tooth which is completely or partially unerupted and is positioned against another tooth, bone or soft tissue so that its further eruption is unlikely, described according to its anatomic position.

Surgical extraction of the impacted mandibular third molars is the most common procedure in oral surgery clinics. Most of the common postoperative complications following lower third molars surgery are pain, trismus and facial swelling. Adequate surgical methods such as selecting an appropriate flap design, minimal bone removal and less trauma to adjacent soft tissues with proper wound closure techniques could decrease the incidence of postoperative sequelae, but not eliminate it.

surgical edema is expected sequel of removal of impacted lower wisdom tooth. Swelling usually reaches at its maximum on 2nd and 3rd postoperatively day and should start reducing by 4th day. Swelling completely resolves by the 7th to 9th day.

Corticosteroids are routinely employed to control the sequelae of inflammation in third molar surgeries. Steroids prevent diapedesis, the initial leakage of fluids from the capillaries, and stabilize the membranes of the cellular lysosomes which hold large quantities of hydrolytic enzymes. There is also a decrease in the formation of bradykinin, a powerful vasodilating substance. Steroids act by suppression of leucocyte and macrophage accumulation at the inflammatory site by interfering with capillary dilatation, fibrin deposition and prevention of prostaglandin synthesis by inhibiting the arachidonic acid cascade.

Trypsin-chymotrypsin is proteolytic enzymes that acts as anti-inflammatory agents. The concentration of enzymes determined as esterase in blood plasma is increased after trypsin chymotrypsin administration. Since the inflammatory process is thought to be due to peptides elaborated at the site of tissue trauma, it has been postulated that the increased blood esterase due to trypsin chymotrypsin administration inhibits inflammation by hydrolytic degradation of the inflammatory peptides.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy patients (ASA I) patient free of any systemic diseases that could interfere with wound healing or surgical operation.
* Free of any recent anti-inflammatory drug intake or being under long term treatment with medicaments that will obscure the assessment of the inflammatory response as NSAIDs, steroids, or antihistamines
* Free from allergy to the drugs used in the study
* Patients requiring surgical removal of the mandibular impacted third molar

Exclusion Criteria:

* Patients who are ASA II to ASA VI.
* Patients already on corticosteroids through any route.
* Patients with known allergy to any drugs.
* Pregnant and lactating females
* Patient not consenting to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
comparison of clinical efficacy of submucosal dexamethasone and oral trypsin-chymotrypsin for reduction of postoperative sequelae after lower third molar surgery | 3 months
  previous study had shown submucosal dexamethasone is more effective than oral trypsin chymotrypsin

CONTACTS AND LOCATIONS:
Locations (1):
- Bp Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Undecided